CLINICAL TRIAL: NCT04686006
Title: Effectiveness of Classical Potassium Iodide Therapy for the Treatment of Untreated Patients With Graves' Hyperthyroidism, Avoiding Thionamide Drugs With Serious Side Effects of Agranulocytosis, Liver Injury, Vasculitis, Embryopathy or Frequent Side Effects of Skin Eruption
Brief Title: Effective Iodide Therapy for Untreated Patients With Graves' Hyperthyroidism Avoiding Thionamide Drugs With Many Side Effects
Status: Completed | Type: Observational
Sponsor: Kyushu University (Other)
Responsible Party: Principal Investigator, Ken Okamura, Professor emeritus, Kyushu University
Other Study IDs: KyushuU Iodide 1
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Graves Disease
MeSH Terms: conditions — Graves Disease | interventions — Potassium Iodide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Graves disease
  Interventions: Drug: Potassium Iodide

INTERVENTIONS:
Drug: Potassium Iodide

SUMMARY:
As the drug treatment of Graves' hyperthyroidism, Plummer reported the effectiveness of excess iodide in 1923 and iodide was used as the therapy for Graves' hyperthyroidism starting from the 1930s. After the introduction of more potent antithyroid drug, thionamide, most thyroidologists preferred to use thionamide expecting potent antithyroid effect, but some careful thyroidologists continued to prescribe iodide in mild type Graves' hyperthyroidism. Recently, American and Europe Thyroid Association recommended methylmercaptoimidazole (MMI), one of the potent thionamide drugs, as the first-choice drug for Graves' hyperthyroidism. However, it became apparent that thionamide has serious side effects such as not only agranulocytosis, but also severe liver injury, MPO-ANCA related vasculitis and embryopathy in the pregnant women. In Japan, one patient died of thionamide-induced agranulocytosis every year. The incidence of side effects including minor side effect of drug eruption is more than 10%. We used to treat the patients with Graves' hyperthyroidism with MMI, as we reported in J Clin Endocrinol Metab 65:719, 1987. However, many side effects of thionamide prompted us to revive the treatment with classical KI in our outpatient clinic and found that KI was effective in the patients who showed side effects to thionamide, resulting in remission (reported in J Clin Endocrinol Metab 99:3995, 2014). Therefore, we began to treat the patients without serious complications such as heart failure or arrhythmia, with 100mg KI since 1996 and followed for 180 days. We were surprised to find that serum thyroid hormone level decreased in all the patients. Thionamide drugs were added only when euthyroidism could not be achieved by KI alone. Compared with thionamide, side effect of KI was almost none. Between 1996 and 2004, about 504 patients were treated with KI and a third of the patients were successfully treated with KI alone and other patients were also successfully treated with the combination of KI and thionamide, suggesting additive effect, or by radioactive iodine therapy. The long term prognosis of the patients initially treated with KI was almost the same as the patients initially treated with MMI. Our clinical experience suggested that patients with Graves' hyperthyroidism are also susceptible to excess iodide, as in the cases with Hashimoto thyroiditis, and this suppressive effect of excess iodide on the thyroid gland is a useful information for many patients suffering from Graves' hyperthyroidism and thionamide side effects.

ELIGIBILITY:
Inclusion Criteria: Untreated Graves' hyperthyroidism. (elevated serum free T4 and/or free T3 level, suppressed serum TSH level, positive anti-TSH receoptor antibody and high thyroidal radioactive iodine uptake -

Exclusion Criteria: dropped out patients within 180 days

-

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 504 (Actual)
Dates: Start 1996-04-01 (Actual); Primary Completion 2005-07-01 (Actual)

PRIMARY OUTCOMES:
Improvement of thyroid function | 180 days
  Normalization of serum free T4 level and TSH level during first 180 days on potassium iodide